CLINICAL TRIAL: NCT05867030
Title: A Phase Ib/III Study to Evaluating the Efficacy and Safety of Parsaclisib in Combination With Rituximab and Lenalidomide Versus Rituximab in Combination With Lenalidomide in Subjects With Relapsed or Refractory Follicular Lymphoma
Brief Title: Parsaclisib in Patients With Relapsed or Refractory Follicular Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development strategy adjustment
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIBI376A301
Record Dates: First submitted 2023-04-10; First posted 2023-05-19 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Lenalidomide; Rituximab; parsaclisib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parsaclisib+rituximab (Experimental): parsaclisib（2.5 mg QD，D1~D14/ per28 days）+rituximab ( 375mg/m2, IV, C1D1\D8\D15\D22, C2D1\C3D1\C4D1\C5D1).
  Interventions: Drug: rituximab; Drug: parsaclisib
- Parsaclisib+rituximab + lenalidomide (Experimental): parsaclisib（2.5 mg QD，D1~D14/ per28 days）+rituximab( 375mg/m2, IV, C1D1\D8\D15\D22, C2D1\C3D1\C4D1\C5D1)+lenalidomide( 20mg PO, D1-D21/Cycle, no more than 12cycles).
  Interventions: Drug: lenalidomide; Drug: rituximab; Drug: parsaclisib

INTERVENTIONS:
Drug: lenalidomide — lenalidomide is administered orally
  Other Names: Lainamei
  Arms: Parsaclisib+rituximab + lenalidomide
Drug: rituximab — rituximab is administered intravenously
  Other Names: Halpryza
Drug: parsaclisib — parsaclisib is administered orally
  Other Names: IBI376

SUMMARY:
A Phase Ib/III, Multicenter, double-blinded study of Parsaclisib, a PI3Kδ Inhibitor, in Patients with Relapsed or Refractory Follicular Lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Histopathological diagnosis as FL Grade1, 2 or 3a
3. The patient is not suitable or refuse the hematopoietic stem cell transplantation(HSCT).
4. Presence of radiographically measurable lymph nodes or extranodal lesions, defined as at least one lesion longest diameter (LD) measurements > 1.5 cm and longest vertical diameter (LPD) measurements ≥1.0 cm.
5. Life expectancy ≥12 weeks.

Exclusion criteria:

1. Known histological transformation of diffuse large B-cell lymphoma (DLBCL) from indolent non-Hodgkin lymphoma (iNHL).
2. A history of central nervous system lymphoma (primary or metastatic) and leptomeninges dease.
3. Previously received Idelalisib, other selective PI3Kδ inhibitors or generic PI3K inhibitor treatment.
4. Previously received Bruton tyrosine kinase inhibitors (e.g., ibrutinib).
5. pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-28 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with a complete response (CR) at the best overall response (BOR) assessed by the investigators (Complete Response Rate , CRR) | within 6 months after last patient enrolled, an average of 2 years
The incidence of treatment-emergent adverse event (TEAE) and the incidence of adverse events of special interest (AESI) leading to permanent discontinuation and/or dose-reduction | within 6 months after last patient enrolled, an average of 2 years
The duration from randomization to disease progression as assessed by an Independent Evaluation Committee (IRC) according to the revised Lymphoma Response Evaluation Criteria (Lugano 2014 criteria) or all-cause death. | up to all subjects reached PFS endpoint, an average of 5 year

SECONDARY OUTCOMES:
The incidence of treatment-emergent adverse event (TEAE) and the incidence of adverse events of special interest (AESI) leading to permanent discontinuation and/or dose-reduction | within 12 months after last patient enrolled, an average of 2.5 years
Percentage of subjects achieving CR or PR in the analysis population evaluated by IRC or investigator according to the Lugano 2014 criteria. | Up to all subjects complete the study treatment, an average of 5 years